CLINICAL TRIAL: NCT04511858
Title: Difference in Central Fatigue During Two Ultra-endurance Practices: Running vs. Cycling
Acronym: FAT-CENTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19CH217; 2020-A01714-35 (Other: ANSM)
Record Dates: First submitted 2020-07-31; First posted 2020-08-13 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Ultra-marathon Runners
Keywords: central fatigue; peripheral fatigue; ultra-endurance exercise; corticospinal excitability

STUDY DESIGN:
Intervention Model Description: Prospective study of physiopathology on subjects specializing in endurance and ultra-endurance: comparing running vs. cycling. Cross-over: each subject will carry out the 2 experimental conditions (running and cycling) according to a randomized order of passage, respecting a wash-out of 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Running endurance (Experimental): Athletes wiil run for 5 hours in a row.
  Interventions: Other: maximum effort test on a treadmill
- Cycling endurance (Experimental): Athletes wiil cycle for 5 hours in a row.
  Interventions: Other: maximum effort test on a cycloergometer

INTERVENTIONS:
Other: maximum effort test on a cycloergometer — 5 h test on cycloergometer
  Arms: Cycling endurance
Other: maximum effort test on a treadmill — 5 h test on treadmill
  Arms: Running endurance

SUMMARY:
The mechanisms contributing to muscle fatigue in extreme long-duration exercise bouts are poorly understood. Ultra-endurance exercise is an excellent model for the study of adaptive responses to extreme loads and stress and it is an especially useful model for documenting the origins of central fatigue. This protocol will compare fatigue during and after ultra-endurance exercise bouts that result in moderate lower-limb tissue damage (i.e. cycling) or significant damage (i.e. running). The results of this protocol will allow us to further understanding of the reasons for major central fatigue, i.e. within the central nervous system, in ultra-endurance.

ELIGIBILITY:
Inclusion Criteria:

* Specialist in endurance and ultra-endurance. in the 2 disciplines: running and cycling (triathletes, duathletes or trailers achieving at least 30% of their training volume in cycling), and having at least finished one long distance event in the last 2 years,
* Affiliated or beneficiary of a social security scheme.
* Signature of the consent form

Exclusion Criteria:

* Any subject who has been injured in the 3 months prior to the protocol
* Anyone with chronic joint pathologies (e.g.: repetitive sprains, patellar or ligament problems).
* Any subject with chronic or central neurological pathologies
* Any subject with a contraindication to magnetic stimulation
* Use of neuro-active substances likely to alter cortico-spinal excitability (hypnotics, antiepileptics, psychotropic drugs, muscle relaxants) on the study.
* Contraindication to the application of a magnetic field:

  * Heart or respiratory insufficiency.
  * Subject with a cardiac pace maker.
  * Cardiac valve wear and serious cardiovascular diseases.
  * Presence of prosthetic material or ferromagnetic foreign bodies in the head.
  * Presence of cochlear implants or ocular prosthetic material.
  * History of neurosurgical interventions.
  * Neurological diseases that may affect brain structures and cognitive abilities (e.g., intracranial tumour, multiple sclerosis, history of stroke or traumatic brain injury).
  * History of comitiality, contralateral knee disease or musculoskeletal disease.
* Any subject participating at the same time in another interventional experiment requiring physical exercise.
* Any subject who has taken corticosteroids within 3 months (inhalation, infiltration or history of prolonged corticosteroid therapy).
* Any subject under guardianship or curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum level of voluntary activation of relative central fatigue | Before and immediately after 5h exercise
  measured in isometric mode of the knee extensors, between the value before and immediately after a 5-hour cycling or running event at the same relative intensity

SECONDARY OUTCOMES:
Maximum level of voluntary activation of fatigue centrale absolute | Before and immediately after 5h exercise
  measured in isometric mode of the knee extensors, between the value before the 5h cycling or running and the value after absolute exhaustion
Maximum level of voluntary activation with electrical evoked activation | Before and immediately after 5h exercise
  tests with measurement of the maximum voluntary with evoked electrical between the value before and immediately after a 5-hour cycling or running event at the same relative intensity
Spinal excitability | Before and immediately after 5h exercise
  thoracic spine stimulation for the recording of thoracic motor evoked potentials
Corticospinal excitability | Before and immediately after 5h exercise
  stimulation of the motor cortex for recording motor evoked potentials
Cortical excitability | Before and immediately after 5h exercise
  ratio between stimulation of the motor cortex and thoracic spine stimulation
Measurement of isometric force values | Before and immediately after 5h exercise
  subjects sitting on a Cybex type seat, with the knee and hip angle set at 90°. The foot will be attached to a strain-gauge sensor using a velcro strap attached to the ankle above the medial malleolus.
Measurement of speed, force and power values | Before and immediately after 5h exercise
  assessment of fatigue in dynamic mode (calculation of the force/speed profile)
Red blood cells | Before and immediately after 5h exercise
  blood sample
Platelets | Before and immediately after 5h exercise
  blood sample
White blood cells | Before and immediately after 5h exercise
  blood sample
Hemoglobin | Before and immediately after 5h exercise
  blood sample
Mean corpuscular hemoglobin concentration | Before and immediately after 5h exercise
  blood sample
C-reactive protein | Before and immediately after 5h exercise
  blood sample
Creatine PhosphoKinase | Before and immediately after 5h exercise
  blood sample
Interleukines | Before and immediately after 5h exercise
  blood sample
Lactate | Before and immediately after 5h exercise
  blood sample
Measurement of the time maintained at the speed corresponding to the 2nd ventilatory threshold | Before and immediately after 5h exercise
  On treadmill
measurement of the time maintained at the power corresponding to the 2nd ventilatory threshold | Before and immediately after 5h exercise
  On Cycloergometer

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Guillaume MILLET, PhD, Study Director — SAINT-ETIENNE UNIVERSITY
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No